CLINICAL TRIAL: NCT02649881
Title: Diagnosis of Macrophage Coronary Plaque by Optical Tomographic Imaging : A Comparative Study With Coronary Artery of the Transplanted or Autopsy Heart
Brief Title: Diagnosis of Macrophage Coronary Plaque by Optical Tomographic Imaging
Acronym: OCT pathology
Status: Completed | Type: Observational
Sponsor: Young-Hak Kim, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Young-Hak Kim, MD, PhD, Division of Cardiology, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2015-03
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Atherosclerotic Plaque
Keywords: macrophage; vulnerable coronary plaque
MeSH Terms: conditions — Plaque, Atherosclerotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- isolated heart from heart transplantation
  Interventions: Procedure: The heart subject will undergo OCT

INTERVENTIONS:
Procedure: The heart subject will undergo OCT

SUMMARY:
This study evaluated optimal macrophage diagnosis algorithm through comparative analysis between coronary artery, OCT image, and IVUS, and improve a diagnosis rate of vulnerable coronary plaque accompanied with macrophage infiltration.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Patients who are to receive heart transplantation
* Patients or their legal representatives who gave a prior written consent

Exclusion Criteria:

* Impossible to OCT and IVUS analysis due to severe coronary stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is targeted at the isolated heart voluntarily donated from adult patients who receive heart transplantation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
ROC curve of diagnosis | within 48 hours
  Receiver Operating Characteristic curve of diagnosis through existing NSD(normalized standard deviation)-based method and developed algorithm in the diagnosis of coronary plaque accompanied with macrophage infiltration

SECONDARY OUTCOMES:
fibrin accumulation | within 48 hours
neoatherosclerosis | within 48 hours
elastic lamia | within 48 hours
cholesterol crystal | within 48 hours
microcalcification | within 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No
This is not publicly funded trial.